CLINICAL TRIAL: NCT06794424
Title: Impact of Ziwig Endotest® on the Decision and Management of Patients with Chronic Disabling Pelvic Pain Strongly Suggestive of Endometriosis and Presenting with a Negative or Uncertain Baseline Imaging Workup
Brief Title: Impact of Ziwig Endotest® on the Management of Patients with Clinical Symptoms of Endometriosis Inconsistent with Their Imaging Work-up
Acronym: ENDOBEST
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ZIWIG (Industry)
Collaborators: Monitoring Force Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ZWG-24-04
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Endometriosis
Keywords: Endometriosis; Endotest; Management of endometriosis; Clinical and radiological discrepancies
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Performing Ziwig Endotest® (Experimental)
  Interventions: Diagnostic Test: Ziwig Endotest®

INTERVENTIONS:
Diagnostic Test: Ziwig Endotest® — Saliva sampling for Endometriosis diagnostic

SUMMARY:
The goal of this study is to evaluate the impact of Ziiwg Endotest on patient management decisions before and after the test. The main questions it aims to answer are:

* Does the test reduce the intention and number of laparoscopies in women whose decision to undergo laparoscopy was made before the test result was obtained?
* Does the test change management decisions in women with no prior indication for diagnostic laparoscopy?

Study will compare the patient management decision before and after the test.

The acts and procedures performed as part of this research are :

* Aa saliva sampling (Ziwig Endotest) at inclusion
* A mutidisciplinary meeting post test (if applicable)
* Completion at inclusion and 6 month of a quality-of-life questionnaire (EHP-5)
* Completion at inclusion and 6 month of a VAS for pain
* Completion at inclusion and 6 month of a Likert satisfaction scale
* A test results Announcement consultation
* A visit at 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Female aged 18 to 43
2. Strong clinical suspicion of endometriosis based on the following suggestive symptoms: chronic pelvic pain (> 6 months) that is suggestive and disabling (ENA ≥ 8, absenteeism or resistance to level 1 analgesics) ± deep dyspareunia or painful hematuria/micturition with menstrual rhythm or painful rectal discharge/defecation with menstrual rhythm.
3. Endovaginal ultrasound and MRI (unless contraindicated, in which case only one of the 2 examinations is required*) less than 1 year old and of sufficient quality , in compliance with the endometriosis protocol recommended by the HAS**.
4. Clinical-radiological discrepancy confirmed by the investigating gynecologist and a referent radiologist at the investigating center, in compliance with the protocol's positivity criteria and the French ENDOVALIRM guidelines (for characterizing deep lesions on MRI) and/or the ESUR 2017 guidelines (for ovarian lesions) and/or the SUR-US 2024 guidelines (for ultrasound).
5. Woman has dated and signed the consent form.
6. Speaks and understands French
7. Affiliated with the French healthcare system

Exclusion Criteria:

1. Endometriosis diagnosed according to imaging protocol positivity criteria
2. Differential diagnosis and/or adenomyosis made
3. History of isolated dysmenorrhea well controlled by hormonal contraception and no immediate desire for pregnancy,
4. Absence of pelvic pain strongly suggestive of endometriosis.
5. Isolated fatigue
6. Aetiological work-up incomplete or pending before deciding on initial medical decision (infertility work-up in progress, waiting for specialist opinion (algologist, psychologist, etc.), waiting for important test results),
7. Infertility work-up (current or previous), with no signs suggestive of endometriosis.
8. Search for recurrence of known endometriosis
9. Laparoscopy for gynecological reasons other than suspected endometriosis
10. History of cancer
11. Pregnant or breast-feeding women
12. Current bacterial or viral infection or less than one month old
13. Participation in an interventional study or in the exclusion period of an interventional study

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2500 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in the number of laparoscopies related to the test result in women whose decision to undergo laparoscopy was made in multidiscplinary meeting before the test result was obtained. MCID 20% | After 6 months visits
  The criterion is estimated after the test result is known.
  Each of these criteria is estimated independently at 3 different times:
  1. After knowledge of the test result, management decided by the physician who carried out the inclusion consultation or at the PCR.
  2. At the end of the consultation, shared decision
  3. At 6 months: by the adjudication committee: positive opinion
  A hierarchical sequential analysis will be carried out independently according to the following scheme:
  Sequence 1: decisional impact of the test on the management decision, if conclusive compared with MCID (main criterion) → sequence 2: decisional impact of the test on the medical decision shared with the patient, if conclusive compared with MCID → sequence 3: percentage of favorable adjudications, conclusive if higher than MCID (highest level of evidence of clinical utility)
Changes in subject management related to Ziwig Endotest® result) in women with no prior indication for diagnostic laparoscopy. MCID 30%. | After 6 months visits
  The criterion is estimated after the test result is known.
  Each of these criteria is estimated independently at 3 different times:
  1. After knowledge of the test result, management decided by the physician who carried out the inclusion consultation or at the PCR.
  2. At the end of the consultation, shared decision
  3. At 6 months: by the adjudication committee: positive opinion
  A hierarchical sequential analysis will be carried out independently according to the following scheme:
  Sequence 1: decisional impact of the test on the management decision, if conclusive compared with MCID (main criterion) → sequence 2: decisional impact of the test on the medical decision shared with the patient, if conclusive compared with MCID → sequence 3: percentage of favorable adjudications, conclusive if higher than MCID (highest level of evidence of clinical utility)

IPD SHARING:
Plan to Share IPD: No